CLINICAL TRIAL: NCT05082909
Title: Addition of Probenecid to Penicillin-V Therapy: an Open Label, Cross-over Study in Healthy Volunteers
Brief Title: Addition of Probenecid to Penicillin-V Therapy
Acronym: ADDPROPEN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21HH6936
Record Dates: First submitted 2021-09-17; First posted 2021-10-19 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Infection, Bacterial
Keywords: Penicillin; Probenecid; Pharmacokinetics
MeSH Terms: conditions — Bacterial Infections | interventions — Probenecid

STUDY DESIGN:
Intervention Model Description: Randomised, cross-over study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penicillin alone (Active Comparator): Penicillin orally at dose of either 250mg, 500mg, 750mg QDS for 36 hours.
  Interventions: Drug: Probenecid
- Penicillin plus probenecid (Experimental): Penicillin orally at dose of either 250mg, 500mg, 750mg QDS for 36 hours.
  PLUS
  Probenecid 500mg QDS for 36 hours.
  Interventions: Drug: Probenecid

INTERVENTIONS:
Drug: Probenecid — Addition of 500mg QDS to oral penicillin.

SUMMARY:
This study aims to build on previous work characterising the PK of penicillin-V to explore the potential impact of probenecid on PK-PD target attainment. Achievement of the aims of this study would provide data to support the design of experimental studies exploring the clinical impact of probenecid on treatment outcomes and also provide a rationale for exploration of probenecid's effects on a larger number of beta-lactam antibiotics.

Hypothesis: Addition of probenecid to oral phenoxymethylpenicillin (penicillin-V) has a clinically relevant effect on pharmacokinetic-pharmacodynamic (PK-PD) target attainment.

DETAILED DESCRIPTION:
Participants will be screened and consented to attend Imperial College Clinical Research Facility (CRF) at Hammersmith Hospital on two study visits, at least 7 days apart. For one visit (randomised), participants will be required to take penicillin-V only. For their other visit, they will take penicillin-V plus probenecid at standard recommended dose. Prior to the study visits, participants may be required to have taken 36-hours of penicillin +/- probenecid, documenting this in a dosing diary. On arrival at the CRF, the participant will take an observed dose of penicillin +/- probenecid. They will undergo blood draw via needle phlebotomy or a cannula (participant choice) at 45 and 180 minutes post the observed. Samples will be spun down and frozen at -80oC. They will subsequently be analysed using an in-house HPLC-MS/MS methodology to determine total and free-unbound drug concentration.

For analysis, data from this study will be pooled with rich PK data from a prior study that assessed plasma concertation of penicillin-V in healthy volunteers. Pmetrics in R will be used to model the data looking to explore the effect of probenecid on clearance of free-penicillin-V. Probability of target attainment for streptococci species will also be estimated to evaluate the potential clinical impact of the addition of probenecid to routine penicillin-V use. Rich PK data for intravenous benzylpenicillin will be used to estimate PK-PD target attainment and PTAs for intravenous formulations, allowing direct comparison of oral and IV regimes.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers (>18 years old).
* Previously taken penicillin-based antibiotics without allergic response.
* Estimated Glomerular Filtration Rate (eGFR) > 90.

Exclusion Criteria:

* Lacking capacity to consent.
* Documented allergy to penicillin, other beta-lactam antibiotics, or probenecid.
* History of G6PD Deficiency.
* Known blood dyscrasias.
* Anaemia (Hb < 12g/dL female, 13g/dL males).
* Abnormal liver function (ALT, AST, ALP or bilirubin > ULN).
* eGFR < 90.
* Pregnant or likely to become pregnant during study period.
* Breastfeeding women.
* Symptoms consistent with active infection.
* History of gout or uric acid kidney stones.
* Taking regular medication that may interact with probenecid including, but not limited to methotrexate, lorazepam, acetaminophen, oral hypoglycaemic medication, sulfa containing drugs, non-steroidal anti-inflammatory drugs.
* History of evidence of any medical, neurological, or psychological condition that would expose the subject to an undue risk of a significant adverse event or interfere with study assessments during the course of the trial as determined by the clinical judgement of the investigator.
* Recent involvement in other research (within prior 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Rawson, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request with appropriate permissions in place.
Supporting Information: Study Protocol, CSR
Time Frame: The protocol will be available from commencement of study. The clinical study report will be published within 12 months of completion of the study.
Access Criteria: Access via the study principle investigator or online publications.

RESULTS

PARTICIPANT FLOW:
Groups:
- Penicillin 250mg QDS THEN Penicillin 250mg QDS Plus Probenecid 500mg QDS: Sequence:
  1. Penicillin orally at dose of 250mg for 36 hours.
  2. Washout period
  3. Penicillin orally at dose of 250mg PLUS probenecid 500mg QDS for 36 hours.
- Penicillin 500mg QDS THEN Penicillin 500mg QDS Plus Probenecid 500mg QDS: Sequence:
  1. Penicillin orally at dose of 500mg for 36 hours.
  2. Washout period
  3. Penicillin orally at dose of 500mg PLUS probenecid 500mg QDS for 36 hours.
- Penicillin 750mg QDS THEN Penicillin 750mg QDS Plus Probenecid 500mg QDS: Sequence:
  1. Penicillin orally at dose of 750mg for 36 hours.
  2. Washout period
  3. Penicillin orally at dose of 750mg PLUS probenecid 500mg QDS for 36 hours.
- Penicillin 250mg QDS Plus Probenecid 500mg QDS THEN Penicillin 250mg QDS.: Sequence:
  1. Penicillin orally at dose of 250mg PLUS probenecid 500mg QDS for 36 hours.
  2. Washout period.
  3. Penicillin orally at dose of 250mg for 36 hours.
- Penicillin 500mg QDS Plus Probenecid 500mg QDS THEN Penicillin 500mg QDS.: Sequence:
  1. Penicillin orally at dose of 500mg PLUS probenecid 500mg QDS for 36 hours.
  2. Washout period.
  3. Penicillin orally at dose of 500mg for 36 hours.
- Penicillin 750mg QDS Plus Probenecid 500mg QDS THEN Penicillin 750mg QDS.: Sequence:
  1. Penicillin orally at dose of 750mg PLUS probenecid 500mg QDS for 36 hours.
  2. Washout period.
  3. Penicillin orally at dose of 750mg for 36 hours.
Period: Overall Study
Arm/Group | Penicillin 250mg QDS THEN Penicillin 250mg QDS Plus Probenecid 500mg QDS | Penicillin 500mg QDS THEN Penicillin 500mg QDS Plus Probenecid 500mg QDS | Penicillin 750mg QDS THEN Penicillin 750mg QDS Plus Probenecid 500mg QDS | Penicillin 250mg QDS Plus Probenecid 500mg QDS THEN Penicillin 250mg QDS. | Penicillin 500mg QDS Plus Probenecid 500mg QDS THEN Penicillin 500mg QDS. | Penicillin 750mg QDS Plus Probenecid 500mg QDS THEN Penicillin 750mg QDS.
Started | 3 | 4 | 4 | 2 | 6 | 2
Completed | 3 | 4 | 3 (One participant withdrawn after randomisation. Was found to be meeting exclusion criteria for the study) | 2 | 6 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant withdrawn after enrolment in Penicillin 750mg QDS THEN Penicillin 750mg QDS plus probenecid 500mg QDS
Groups:
- Penicillin 250mg QDS THEN Penicillin 250mg QDS Plus Probenecid 500mg QDS: Sequence:
  1. Penicillin orally at dose of 250mg QDS for 36 hours.
  2. Washout period
  3. Penicillin orally at dose of 250mg QDS and probenecid 500mg QDS to oral penicillin for 36 hours.
- Penicillin 500mg QDS THEN Penicillin 500mg QDS Plus Probenecid 500mg QDS: Sequence:
  1. Penicillin orally at dose of 500mg QDS for 36 hours.
  2. Washout period
  3. Penicillin orally at dose of 500mg QDS and probenecid 500mg QDS to oral penicillin for 36 hours.
- Penicillin 750mg QDS THEN Penicillin 750mg QDS Plus Probenecid 500mg QDS: Sequence:
  1. Penicillin orally at dose of 750mg QDS for 36 hours.
  2. Washout period
  3. Penicillin orally at dose of 750mg QDS and probenecid 500mg QDS to oral penicillin for 36 hours
- Penicillin 250mg QDS Plus Probenecid 500mg QDS THEN Penicillin 250mg QDS: Sequence:
  1. Penicillin orally at dose of 250mg QDS and probenecid 500mg QDS to oral penicillin for 36 hours
  2. Washout period
  3. Penicillin orally at dose of 250mg QDS for 36 hours.
- Penicillin 500mg QDS Plus Probenecid 500mg QDS THEN Penicillin 500mg QDS: Sequence:
  1. Penicillin orally at dose of 500mg QDS and probenecid 500mg QDS to oral penicillin for 36 hours
  2. Washout period
  3. Penicillin orally at dose of 500mg QDS for 36 hours.
- Penicillin 750mg QDS Plus Probenecid 500mg QDS THEN Penicillin 750mg QDS: Sequence:
  1. Penicillin orally at dose of 750mg QDS and probenecid 500mg QDS to oral penicillin for 36 hours
  2. Washout period
  3. Penicillin orally at dose of 750mg QDS for 36 hours.
- Total: Total of all reporting groups
Arm/Group | Penicillin 250mg QDS THEN Penicillin 250mg QDS Plus Probenecid 500mg QDS | Penicillin 500mg QDS THEN Penicillin 500mg QDS Plus Probenecid 500mg QDS | Penicillin 750mg QDS THEN Penicillin 750mg QDS Plus Probenecid 500mg QDS | Penicillin 250mg QDS Plus Probenecid 500mg QDS THEN Penicillin 250mg QDS | Penicillin 500mg QDS Plus Probenecid 500mg QDS THEN Penicillin 500mg QDS | Penicillin 750mg QDS Plus Probenecid 500mg QDS THEN Penicillin 750mg QDS | Total
Number analyzed (Participants) | 3 | 4 | 4 | 2 | 6 | 2 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (18) | 55 (11) | 52 (14) | 48 (22) | 67 (6) | 30 (2) | 53 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4 | 0 | 8
  Male | 2 | 3 | 3 | 1 | 2 | 2 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 | 4 | 4 | 2 | 6 | 2 | 21
Weight [Mean (Standard Deviation); unit: Kilograms] | 68 (5) | 68 (8) | 74 (11) | 70 (0) | 71 (6) | 88 (1) | 72 (9)
Height [Mean (Standard Deviation); unit: cm] | 167 (10) | 169 (10) | 170 (5) | 171 (5) | 174 (4) | 179 (3) | 171.5 (7.8)
Creatinine [Mean (Standard Deviation); unit: micromol/L] | 62 (5) | 68 (6) | 69 (2) | 64 (3) | 70 (7) | 78 (5) | 68 (9)
Albumin [Mean (Standard Deviation); unit: g/L] | 42 (3) | 41 (2) | 41 (2) | 41 (3) | 40 (2) | 43 (1) | 41 (2)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Total and Unbound Penicillin-V Concentration
Description: Measurement of blood concentration at 45 minutes post dose with and without probenecid.
Time Frame: 45 minutes post an observed dose.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- 250mg Penicillin Arm 1: Penicillin 250mg QDS THEN Penicillin 250mg QDS Plus Probenecid 500mg QDS
- 250mg Penicillin Arm 2: Penicillin 250mg QDS Plus Probenecid 500mg QDS THEN Penicillin 250mg QDS
- 500mg Penicillin Arm 1: Penicillin 500mg QDS THEN Penicillin 500mg QDS Plus Probenecid 500mg QDS
- 500mg Penicillin Arm 2: Penicillin 500mg QDS Plus Probenecid 500mg QDS THEN Penicillin 500mg QDS
- 750mg Penicillin Arm 1: Penicillin 750mg QDS THEN Penicillin 750mg QDS Plus Probenecid 500mg QDS
- 750mg Penicillin Arm 2: Penicillin 750mg QDS Plus Probenecid 500mg QDS THEN Penicillin 750mg QDS
Arm/Group | 250mg Penicillin Arm 1 | 250mg Penicillin Arm 2 | 500mg Penicillin Arm 1 | 500mg Penicillin Arm 2 | 750mg Penicillin Arm 1 | 750mg Penicillin Arm 2
Number analyzed (Participants) | 3 | 2 | 4 | 6 | 3 | 2
mg/L
  Total penicillin concentration (mg/L) - penicillin alone | 2.07 (0.16) | 2.8 (0.10) | 5.03 (1.46) | 3.62 (1.56) | 6.53 (5.38) | 6.2 (0.8)
  Unbound penicillin concentration (mg/L) - penicillin alone | 0.39 (0.04) | 0.56 (0.01) | 0.97 (0.22) | 0.65 (0.27) | 1.22 (0.34) | 1.08 (0.15)
  Total penicillin concentration (mg/L) - penicillin plus probenecid | 4.83 (0.91) | 7.45 (1.05) | 10.88 (2.41) | 6.50 (3.20) | 12 (2.27) | 12 (3)
  Unbound penicillin concentration (mg/L) - penicillin plus probenecid | 1.58 (0.87) | 1.74 (0.14) | 2.36 (0.59) | 1.52 (0.76) | 2.63 (0.64) | 2.84 (0.77)

2. Primary Outcome: Measurement of Total and Unbound Penicillin-V Concentration
Description: Measurement of blood concentration at 180 minutes post dose with and without probenecid.
Time Frame: 180 minutes post an observed dose.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 250mg Penicillin Arm 1 | 250mg Penicillin Arm 2 | 500mg Penicillin Arm 1 | 500mg Penicillin Arm 2 | 750mg Penicillin Arm 1 | 750mg Penicillin Arm 2
Number analyzed (Participants) | 3 | 2 | 4 | 6 | 3 | 2
mg/L
  Total penicillin concentration (mg/L) - penicillin alone | 0.13 (0.05) | 0.85 (0.45) | 0.98 (0.76) | 0.85 (0.26) | 1.97 (0.76) | 0.45 (0.15)
  Unbound penicillin concentration (mg/L) - penicillin alone | 0.03 (0.01) | 0.15 (0.07) | 0.18 (0.14) | 0.16 (0.05) | 0.35 (0.13) | 0.09 (0.03)
  Total penicillin concentration (mg/L) - penicillin plus probenecid | 1.58 (0.87) | 2.35 (1.15) | 5.18 (2.15) | 2.22 (0.56) | 6.67 (3.09) | 3.55 (1.45)
  Unbound penicillin concentration (mg/L) - penicillin plus probenecid | 0.33 (0.16) | 0.49 (0.21) | 1.18 (0.51) | 0.49 (0.11) | 1.46 (0.78) | 0.81 (0.34)

3. Secondary Outcome: Measurement of Total and Unbound Probenecid Concentration
Description: Measurement of blood concentration at 45 minutes post observed probenecid dose.
  Combined data for all participants given that the same dose of probenecid was taken by all participants.
Time Frame: 45 minutes post an observed dose.
Population: All 20 participants received the same dose (500mg QDS) of probenecid regardless of study arm. Results are therefore presented for all participants for this outcome.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Total Probenecid Concentration; Unbound Probenecid Concentraion: All 20 participants from probenecid 500mg QDS arm of cross-over study.
Arm/Group | Total Probenecid Concentration | Unbound Probenecid Concentraion
Number analyzed (Participants) | 20 | 20
mg/L | 79.0 (21.4) | 6.6 (1.5)

4. Secondary Outcome: Measurement of Total and Unbound Probenecid Concentration
Description: Measurement of blood concentration at 180 minutes post observed probenecid dose.
  Combined data for all participants given that the same dose of probenecid was taken by all participants.
Time Frame: 180 minutes post an observed dose.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Total Probenecid Concentration | Unbound Probenecid Concentraion
Number analyzed (Participants) | 20 | 20
mg/L | 81.1 (20.6) | 6.6 (1.5)

ADVERSE EVENTS:
Time Frame: Data collected over 3 weeks from participant enrolment to final visit completion per participant.
Description: Results have been reported as per our protocol. Results are not reported per arm/group as dose dependent adverse events were not assessed. Assessment of adverse events aimed to compare penicillin alone against penicillin with probenecid, as is presented in this table.
Groups:
- Penicillin Alone: Penicillin orally QDS for 36 hours.
  This data has been grouped to present a comparison of penicillin vs. probenecid irrespective of dose.
- Penicillin Plus Probenecid: Penicillin orally for 36 hours.
  PLUS
  Probenecid 500mg QDS for 36 hours.
  This data has been grouped to present a comparison of penicillin vs. probenecid irrespective of dose.
Arm/Group | Penicillin Alone | Penicillin Plus Probenecid
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 8/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Penicillin Alone (N=20) | Penicillin Plus Probenecid (N=20)
Mild, expected (GI side effects) (Gastrointestinal disorders) | 3 (4) | 5 (7)
Mild, expected (headache) (Nervous system disorders) | 1 (1) | 3 (3)
Unexpected, not related to IMP (Infections and infestations) | 1 (1) | 0 (0) — Flu-like illness
Unexpected, not related to IMP (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Leg pain
Unexpected, possible association with IMP (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Flushing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT05082909/Prot_SAP_000.pdf